CLINICAL TRIAL: NCT00048373
Title: Treatment of Resistant Langerhans Cell Histiocytosis With Etanercept (ENBREL, IMMUNEX, SEATTLE)
Brief Title: Treatment of Resistant Langerhans Cell Histiocytosis With ENBREL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Kenneth McClain, Professor, Pediatrics-Oncology, Baylor College of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H10339; Etanercept
Record Dates: First submitted 2002-10-30; First posted 2002-11-01 (Estimated); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Histiocytosis, Langerhans-Cell
Keywords: LANGERHANS; HISTIOCYTOSIS
MeSH Terms: conditions — Histiocytosis, Langerhans-Cell; Histiocytosis | interventions — Etanercept

INTERVENTIONS:
Drug: Etanercept

SUMMARY:
The purpose of this study is to learn about the response of Langerhans cell histiocytosis (LCH) to Enbrel in patients who have failed to respond to standard therapies. We are also looking specifically at what side effects Enbrel has on patients. We expect to enroll 20 patients on this study and anticipate the subjects active participation to last up to one year.

DETAILED DESCRIPTION:
After subjects have completed the pretreatment evaluations, they will receive an injection of Enbrel - the study drug -(given under the skin) twice weekly. If the subjects disease stabilizes or regresses, they may continue to receive treatment for up to 1 year.

Subjects with disease involvement of risk organs (this means patients have disease in their liver, lung, spleen, or bone marrow): will be admitted to the hospital for observation during the first week of administration of Enbrel. If after the first two doses there appears to be no problems, subjects may be followed as an outpatient with twice weekly evaluation visits (similar to those performed before treatment began) until abnormal blood tests have become normal. Then the frequency of clinic visits will decrease and be similar to those described below for subjects without disease involvement of risk organs.

Subjects without disease involvement of risk organs will be treated as an outpatient. While receiving the treatment, subjects may not receive any other chemotherapy agents. Doctors will be monitoring subjects closely for side effects. Most side effects usually disappear after the treatment is stopped. In the meantime, however, the doctor may prescribe medication to keep these side effects under control.

ELIGIBILITY:
INCLUSION:

* Age: Patients of any age greater than 1 year and up to 65 years of age. An internal medicine board-certified physician will also evaluate adult patients.
* Histologic diagnosis: Patients must have a histologically confirmed LCH that is refractory to standard therapy.
* Recovery from prior therapy: Patients must have recovered from the toxic effects of all prior therapy but may have abnormal hematologic, hepatic, or other lab values secondary to the disease.
* Life expectancy: Patients must have a life expectancy of at least 8 weeks.
* Performance status: Patients must have a Lansky performance status greater than 40 or Karnofsky status greater than 40.
* Informed consent: All patients or their legal guardians (if the patient is < 18 years of age) must sign a document of informed consent indicating their awareness of the investigational nature and the risks of this study. When appropriate the patient will be included in all discussions in order to obtain verbal consent.
* Hematologic status: Patients of any hematologic status may be enrolled since resistant LCH may require considerable transfusion support.
* Durable Power of Attorney (DPA): A DPA must be offered to all patients 18 years of age or older.

EXCLUSION:

* Women of childbearing potential who are pregnant or lactating are excluded.
* Patients with active infections must be treated prior to entry.
* Significant other diseases that the investigator feels will complicate review/evaluation of the study data (example: uncontrolled diabetes, multiple sclerosis).

Ages: 1 Day to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20
Dates: Start 2001-10; Study Completion 2004-04

PRIMARY OUTCOMES:
Response of Langerhans cell histiocytosis

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth McClain, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States